CLINICAL TRIAL: NCT02807181
Title: Prospective, Multicenter, Randomized, Controlled Study Evaluating SIR-Spheres Y-90 Resin Microspheres Preceding Cisplatin-gemcitabine (CIS-GEM) Chemotherapy Versus CIS-GEM Chemotherapy Alone as First-line Treatment of Patients With Unresectable Intrahepatic Cholangiocarcinoma
Brief Title: SIRT Followed by CIS-GEM Chemotherapy Versus CIS-GEM Chemotherapy Alone as 1st Line Treatment of Patients With Unresectable Intrahepatic Cholangiocarcinoma
Acronym: SIRCCA
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Sirtex Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STX0115
Record Dates: First submitted 2016-05-13; First posted 2016-06-21 (Estimated); Results first posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-04

CONDITIONS: Intrahepatic Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Chemotherapy (Cisplatin-Gemcitabine) (Active Comparator): Cisplatin 25mg/m2 in 1000ml 0.9% saline given over 1 hour followed by 500 ml 0.9% saline over 30 minutes, followed by Gemcitabine 1000 mg/m2 in 250-500 ml 0.9% saline over 30 minutes by intravenous infusions on days 1, and 8 of a 21-day cycle.
  Interventions: Drug: Cisplatin-gemcitabine
- Radiation: SIRT + chemotherapy (Cisplatin-Gemcitabine) (Experimental): A single treatment of hepatic arterial injection of SIR-Spheres Y-90 resin microspheres (SIRT) followed 14-16 days later by systemic chemotherapy (ABC-02 CIS-GEM protocol) with an intention to treat with 8 cycles of cisplatin + gemcitabine, or until progression, toxicity or patient choice. Treatment may be continued beyond 8 cycles in the absence of significant disease progression, at the treating clinicians' discretion.
  Interventions: Drug: Cisplatin-gemcitabine; Device: Radiation: SIRT + chemotherapy (cisplatin-gemcitabine)

INTERVENTIONS:
Drug: Cisplatin-gemcitabine — Systemic chemotherapy
  Other Names: CIS-GEM
Device: Radiation: SIRT + chemotherapy (cisplatin-gemcitabine) — SIR-Spheres microspheres followed by systemic chemotherapy
  Arms: Radiation: SIRT + chemotherapy (Cisplatin-Gemcitabine)

SUMMARY:
The study planned to evaluate the benefit of applying Selective Internal Radiation Therapy (SIRT) using SIR-Spheres Y-90 resin microspheres prior to receiving systemic chemotherapy treatment (cisplatin-gemcitabine, or CIS-GEM) in patients with unresectable intrahepatic cholangiocarcinoma. Half of the patients were randomized to CIS-GEM chemotherapy plus SIRT, and half of the patients were randomized to CIS-GEM alone.

DETAILED DESCRIPTION:
This clinical study was a prospective, multicenter, randomized, controlled study evaluating SIR-Spheres Y-90 resin microspheres followed by cisplatin-gemcitabine (CIS-GEM) chemotherapy vs. CIS-GEM chemotherapy alone as first-line treatment of patients with unresectable intrahepatic cholangiocarcinoma.

Randomized patients were to be followed until death, withdrawal of consent, or until end of study.

ELIGIBILITY:
Inclusion Criteria:

* Willing, able and mentally competent to provide written informed consent.
* Aged 18 years or older.
* Histologically or cytologically confirmed unresectable and non-ablatable intrahepatic cholangiocarcinoma.
* Liver-only or liver predominant intrahepatic cholangiocarcinoma. Patient are permitted to have loco-regional lymph node involvement defined as: portal LN </= to 2 cm and/or para aortic LN </= to 1.5 cm in longest diameter, and/or up to 2 indeterminate lung lesions < 1 cm if these lung lesions are positron emission tomography (PET) negative.
* Chemotherapy naïve. Adjuvant chemotherapy is not permitted.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
* Adequate hematological function defined as:

Hemoglobin >/= 10g/dL White Blood Cell count (WBC) >/= 3.0 x 10^9/L Absolute neutrophil count (ANC) >/= 1.5 x 10^9/L Platelet count >/= 100,000/mm^3 - Adequate liver function defined as: Total bilirubin </= 30 umol/L (1.75 mg/dL) Albumin >/= 30 g/L

- Adequate renal function defined as: Serum urea and serum creatinine < 1.5 times upper limit of normal (ULN) Creatinine clearance >/= 45 ml/min (calculated with Cockcroft-Gault Equation)

* Life expectancy of at least 3 months without any active treatment
* Female patients must either be postmenopausal, sterile (surgically or radiation- or chemically-induced), or if sexually active use an acceptable method of contraception during the study.
* Male patients must be surgically sterile or if sexually active must use an acceptable method of contraception during the study.
* Considered suitable to receive either regimen in the clinical judgement of the treating investigator.

Exclusion Criteria:

* Patients with only non-measurable lesions in the liver according to RECIST criteria
* Incomplete recovery from previous liver surgery, e.g. unresolved biliary tree obstruction or biliary sepsis or inadequate liver function
* Biliary stent in situ
* Main trunk Portal Vein Thrombosis (PVT)
* Ascites, even if controlled with diuretics. (A minor peri-hepatic rim of ascites detected at imaging is acceptable).
* Mixed hepatocellular carcinoma - intrahepatic cholangiocarcinoma (HCC-ICC) disease
* History of prior malignancy. Exceptions include in-situ carcinoma of the cervix treated by cone-biopsy/resection, non-metastatic basal and/or squamous cell carcinomas of the skin, recurrent intra-hepatic cholangiocarcinoma post local treatment or any early stage (stage 1) malignancy adequately resected with curative intent at least 5 years prior to study entry
* Suspicion of any bone metastasis/metastases or central nervous system metastasis/metastases on clinical or imaging examination.
* Prior internal or external radiation delivered to the liver.
* Pregnancy; breast feeding.
* Participation within 28 days prior to randomization, in an active part of another clinical study that would compromise any of the endpoints of the study.
* Evidence of ongoing active infection that may affect treatment feasibility or outcome.
* Prior Whipple's procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2017-02-14 (Actual); Primary Completion 2021-04-29 (Actual); Study Completion 2021-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jordi Bruix, MD, Principal Investigator — Head of the Hepatic Oncology Unit, Hospital Clinic; Harpreet Wasan, MD, Principal Investigator — Imperial College Healthcare Hammersmith Hospital
Locations (23):
- Providence Health Care, Spokane, Washington, United States
- Australia (2):
  - Macquarie University Hospital, North Ryde, New South Wales
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
- Cliniques Universitaires Saint-Luc, Brussels, Belgium
- France (11):
  - Hopital Beaujon, Clichy
  - CHU Dijon, Dijon
  - CHU de Grenoble, Grenoble
  - CHU Lyon - Hospital de la Croix-Rousse, Lyon
  - Institut Paoli Calmettes, Marseille
  - CHU Montpellier, Montpellier
  - CHU Nice - Hopital l'Archet 2, Nice
  - Hopital Haut-Leveque, Pessac
  - CHU de Poitiers, Poitiers
  - Centre Eugene Marquis Hospital de Jour, Rennes
  - Hopital Paul Brousse, Villejuif
- U.O. Oncologia Medica 2 Universitaria, Pisa, Italy
- AMC Academic Medical Center, Amsterdam, Netherlands
- Spain (2):
  - Hospital Clinic Barcelona, Barcelona
  - Clinica Universitaria de Navarra, Pamplona
- United Kingdom (4):
  - Hammersmith Hospital Imperial College Healthcare NHS Trust, London
  - The Christie NHS Foundation Trust, Manchester
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Metropolitan Borough of Wirral
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Chemotherapy (Cisplatin-Gemcitabine) | Radiation: SIRT + Chemotherapy (Cisplatin-Gemcitabine)
Started | 48 (randomized population) | 41 (randomized population)
Completed | 11 | 9
Not Completed | 37 | 32
Not completed — Death | 28 | 24
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 0 | 2
Not completed — Subject decision | 1 | 0
Not completed — Biopsy of tumor removed from resection | 1 | 0
Not completed — In Study | 3 | 3
Not completed — Post Progression | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chemotherapy (Cisplatin-Gemcitabine) | Radiation: SIRT + Chemotherapy (Cisplatin-Gemcitabine) | Total
Number analyzed (Participants) | 48 | 41 | 89
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 14 | 38
  >=65 years | 24 | 27 | 51
Age, Continuous [Mean (Full Range); unit: years] | 61.94 [29 to 81] | 67.17 [46 to 88] | 64.35 [29 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 23 | 45
  Male | 26 | 18 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 16 | 10 | 26
  Unknown or Not Reported | 30 | 30 | 60
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 15 | 9 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 32 | 31 | 63
Region of Enrollment [Number; unit: participants]
  Netherlands | 2 | 3 | 5
  Belgium | 4 | 0 | 4
  United States | 1 | 0 | 1
  Italy | 1 | 0 | 1
  United Kingdom | 5 | 4 | 9
  Australia | 1 | 2 | 3
  France | 30 | 30 | 60
  Spain | 4 | 2 | 6
Extra-hepatic disease [Count of Participants; unit: Participants]
  Present | 20 | 20 | 40
  Absent | 28 | 21 | 49
ECOG Performance Scale [Count of Participants; unit: Participants] — Eastern cooperative oncology group (ECOG) performance status 0 versus 1 as per the study inclusion criterion. 0=Fully active, able to carry on all pre-disease performance without restriction; 1=Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g. light housework, office work.
  Participants
    0 | 33 | 33 | 66
    1 | 15 | 8 | 23
Cirrhosis [Count of Participants; unit: Participants]
  Present | 7 | 4 | 11
  Absent | 41 | 37 | 78
Extent of liver involvement [Count of Participants; unit: Participants]
  Non-whole | 32 | 30 | 62
  Whole | 16 | 11 | 27
Prior Treatment [Count of Participants; unit: Participants]
  Yes | 35 | 26 | 61
  No | 13 | 15 | 28

OUTCOME MEASURES:

1. Primary Outcome: Survival at 18 Months
Description: Survival at 18 months is defined as the proportion of patients still alive 18 months from the date of randomization. The outcome was analyzed but the clinical database is not deemed to be reliable.
Time Frame: 18 months following the date of randomization.
Population: Randomized Population
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy (Cisplatin-Gemcitabine) | Radiation: SIRT + Chemotherapy (Cisplatin-Gemcitabine)
Number analyzed (Participants) | 48 | 41
Participants
  Yes | 25 | 23
  No | 23 | 18

2. Secondary Outcome: Liver-specific Progression Free Survival (PFS)
Description: Liver-specific PFS was defined as the number of days between randomization and the date of first tumor progression in the liver. Diagnosis of tumor progression was to be made using RECIST 1.1.
Time Frame: From date of randomization to the first documented date of progression in the liver or date of death from any cause, assessed up to 36 months..
Population: The data set we received for analysis showed only 17 CIS-GEM participants and 16 SIRT+CIS GEM participants with reported liver tumor progression data available. Due to database issues, the validity and reliability of this data is not complete.
Measure: Mean (Full Range); unit: Days to first tumor progression
Arm/Group | Chemotherapy (Cisplatin-Gemcitabine) | Radiation: SIRT + Chemotherapy (Cisplatin-Gemcitabine)
Number analyzed (Participants) | 17 | 16
Days to first tumor progression | 323 [82 to 712] | 369 [102 to 875]

3. Secondary Outcome: Progression Free Survival (PFS) at Any Site
Description: PFS was defined as the time interval between randomization and the date of tumor progression. Diagnosis of tumor progression was to be made using RECIST 1.1. The outcome was not analyzed due to unreliability of the clinical database.
Time Frame: From date of randomization to the date of progression at any site until the first date of documented tumor progression at any site or date of death from any cause, assessed up to 36 months.
Population: The data set we received for analysis showed 38 CIS-GEM participants and 27 SIRT+CIS GEM participants with reported tumor progression data available for any site. Due to database issues, the validity and reliability of this data is not complete
Measure: Mean (Full Range); unit: Days to tumor progression
Arm/Group | Chemotherapy (Cisplatin-Gemcitabine) | Radiation: SIRT + Chemotherapy (Cisplatin-Gemcitabine)
Number analyzed (Participants) | 38 | 27
Days to tumor progression | 332 [40 to 712] | 424 [102 to 875]

4. Secondary Outcome: Objective Response Rate by RECIST 1.1 and Refined RECIST - Liver
Description: The outcome was not analyzed due to unreliability of the clinical database.
Time Frame: From the date of first treatment until the date of date of first documented progression in the liver, assessed up to 36 months.
Population: The data we received showed 85 of our 89 subjects with any RECIST data present. These data were not available nor complete for each visit due to early study termination and database issues. Any available data is reflected in the table. The validity and reliability of these data are not complete.
Measure: Count of Units; unit: Number of Responses (RECIST 1.1+RRECIST)
Units Other Than Participants: Number of Responses (RECIST 1.1+RRECIST)
Groups:
- Chemotherapy (Cisplatin-Gemcitabine) Total Subjects: Cisplatin 25mg/m2 in 1000ml 0.9% saline given over 1 hour followed by 500 ml 0.9% saline over 30 minutes, followed by Gemcitabine 1000 mg/m2 in 250-500 ml 0.9% saline over 30 minutes by intravenous infusions on days 1, and 8 of a 21-day cycle.
  Cisplatin-gemcitabine: Systemic chemotherapy
Arm/Group | Chemotherapy (Cisplatin-Gemcitabine) Total Subjects | Radiation: SIRT + Chemotherapy (Cisplatin-Gemcitabine)
Number analyzed (Participants) | 44 | 41
Number analyzed (Number of Responses (RECIST 1.1+RRECIST)) | 396 | 416
Number of Responses (RECIST 1.1+RRECIST)
  Complete Response (CR) : RECIST 1.1 | 22 | 10
  Complete Response (CR) : Refined RECIST | 21 | 10
  Partial Response (PR) : RECIST 1.1 | 25 | 58
  Partial Response (PR) : Refined RECIST | 24 | 56
  Progressive Disease (PD) : RECIST 1.1 | 23 | 13
  Progressive Disease (PD) : Refined RECIST | 22 | 13
  Stable Disease (SD) : RECIST 1.1 | 113 | 110
  Stable Disease (SD) : Refined RECIST | 105 | 105
  Not Evaluable : RECIST 1.1 | 13 | 8
  Not Evaluable : Refined RECIST | 13 | 8
  Incomplete Form : RECIST 1.1 | 2 | 9
  Incomplete Form : Refined RECIST | 13 | 16

5. Secondary Outcome: Objective Response Rate by RECIST 1.1 and Refined RECIST - at Any Site
Description: The outcome was not analyzed due to unreliability of the clinical database.
Time Frame: From the date of first treatment until progression at any site, assessed up to 36 months.
Population: as for outcome 4
Measure: Count of Units; unit: Number of Responses (RECIST 1.1+RRECIST)
Units Other Than Participants: Number of Responses (RECIST 1.1+RRECIST)
Arm/Group | Chemotherapy (Cisplatin-Gemcitabine) | Radiation: SIRT + Chemotherapy (Cisplatin-Gemcitabine)
Number analyzed (Participants) | 44 | 41
Number analyzed (Number of Responses (RECIST 1.1+RRECIST)) | 396 | 416
Number of Responses (RECIST 1.1+RRECIST)
  Complete Response (CR) : RECIST 1.1 | 22 | 8
  Complete Response (CR) : Refined RECIST | 22 | 7
  Partial Response (PR) : RECIST 1.1 | 28 | 28
  Partial Response (PR) : Refined RECIST | 27 | 48
  Progressive Disease (PD) : RECIST 1.1 | 42 | 42
  Progressive Disease (PD) : Refined RECIST | 38 | 34
  Stable Disease (SD) : RECIST 1.1 | 103 | 102
  Stable Disease (SD) : Refined RECIST | 98 | 96
  Not Evaluable : RECIST 1.1 | 1 | 7
  Not Evaluable : Refined RECIST | 0 | 7
  Incomplete Form : RECIST 1.1 | 2 | 9
  Incomplete Form : Refined RECIST | 13 | 16

6. Secondary Outcome: Overall Survival
Description: The outcome was not analyzed due to unreliability of the clinical database.
Time Frame: From date of randomization until the date of death from any cause, assessed up to 36 months.
Population: Overall survival data assessed until 36 months can be calculated for 42 CIS GEM participants and 36 SIRT+CIS GEM participants due to early termination and database errors. The validity and reliability of these data are not complete.
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy (Cisplatin-Gemcitabine) | Radiation: SIRT + Chemotherapy (Cisplatin-Gemcitabine)
Number analyzed (Participants) | 42 | 36
Participants
  Number of Participants Alive | 14 | 12
  Number of Participants Expired | 28 | 24

7. Secondary Outcome: Liver Surgical Resection and Ablation Rate
Description: To assess the number of patients in each arm who are downstaged by protocol therapy and can proceed to liver resection or ablation. The specific assessments will be the classification of resection as R0, R1 or R2, the presence of viable tumor or fibrosis, and the nearest resection margin. The outcome was not analyzed due to unreliability of the clinical database.
Time Frame: 18 months following the date of randomization.
Population: Data were collected for only 14 unique patients within the study due to early study termination and database issues. Any available data are reflected in the table. The validity and reliability of these data are not complete.
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy (Cisplatin-Gemcitabine) | Radiation: SIRT + Chemotherapy (Cisplatin-Gemcitabine)
Number analyzed (Participants) | 7 | 7
Participants
  Count of participants with resection only | 4 | 4
  Count of participants with resection and ablation | 1 | 1
  Count of participants with no resection or ablation | 2 | 2

8. Secondary Outcome: Incidence of Adverse Events (Safety and Tolerability)
Description: Adverse events (AEs) as assessed by CTCAE v. 4.0. Summaries of non-serious AEs (clinical database, MedDRA 20.1) and serious adverse events (SAEs; pharmacovigilance database, MedDRA 25.1) are provided for information only in the 'Adverse Events' section - the data are deemed unreliable.
Time Frame: Informed consent until 28 days post last dose of protocol chemotherapy.
Population: The following endpoints reflects safety and tolerability data related to Adverse Event grade by category. Counts of participants with Grade 3 or higher adverse event severity by AE category by treatment arm are shown below.
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy (Cisplatin-Gemcitabine) | Radiation: SIRT + Chemotherapy (Cisplatin-Gemcitabine)
Number analyzed (Participants) | 48 | 41
Participants
  Serious Adverse Events | 17 | 20
  Grade 3 or higher Blood and lymphatic system disorders | 15 | 16
  Grade 3 or higher Cardiac disorders | 2 | 2
  Grade 3 or higher Gastrointestinal disorders | 5 | 5
  Grade 3 or higher General disorders and administration site conditions | 5 | 8
  Grade 3 or higher Hepatobiliary disorders | 3 | 4
  Grade 3 or higher Immune system disorders | 0 | 1
  Grade 3 or higher Infections and infestations | 3 | 0
  Grade 3 or higher Injury, poisoning and procedural complications | 0 | 1
  Grade 3 or higher Investigations | 16 | 26
  Grade 3 or higher Metabolism and nutrition disorders | 3 | 4
  Grade 3 or higher Musculoskeletal and connective tissue disorders | 0 | 1
  Grade 3 or higher Nervous system disorders | 0 | 3
  Grade 3 or higher Psychiatric disorders | 0 | 1
  Grade 3 or higher Renal and urinary disorders | 2 | 0
  Grade 3 or higher Reproductive system and breast disorders | 1 | 0
  Grade 3 or higher Respiratory, thoracic and mediastinal disorders | 4 | 1
  Grade 3 or higher Skin and subcutaneous tissue disorders | 0 | 1
  Grade 3 or higher Surgical and medical procedures | 0 | 2
  Grade 3 or higher Vascular disorders | 4 | 4

ADVERSE EVENTS:
Time Frame: Up to 3.6 years
Description: AEs from time of informed consent up to 28 days post last dose of chemo, and any treatment-related (TR) AEs at any time were recorded. SAEs and TR AEs were followed until resolution, death, or end of study. Per protocol, disease progression events were not considered AEs, but lack of efficacy. If any disease progression events occurred, no data was collected, and they were not documented in the database. All recorded AEs that met the Results Data Element Definitions were reported.
Arm/Group | Chemotherapy (Cisplatin-Gemcitabine) | Radiation: SIRT + Chemotherapy (Cisplatin-Gemcitabine)
All-Cause Mortality (participants affected / at risk) | 28/48 | 24/41
Serious Adverse Events (participants affected / at risk) | 17/48 | 21/41
Other Adverse Events (participants affected / at risk) | 47/48 | 41/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemotherapy (Cisplatin-Gemcitabine) (N=48) | Radiation: SIRT + Chemotherapy (Cisplatin-Gemcitabine) (N=41)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (4) | 0 (0)
Aortic valve disease (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (3) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (2) | 2 (2)
Diaphragmatic hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemoperitoneum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Spigelian hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)
Chills (General disorders) | 1 (1) | 0 (0)
Condition aggravated (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 4 (5)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Strangulated hernia (General disorders) | 1 (1) | 0 (0)
Haemobilia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic pain (Hepatobiliary disorders) | 0 (0) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Campylobacter infection (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Pneumocytis jirovecii pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post embolization syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural shock (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radiation hepatitis (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 2 (2)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Posterior reversable encephalopathy syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Aortic valve replacement (Surgical and medical procedures) | 0 (0) | 1 (1)
Drug delivery device placement (Surgical and medical procedures) | 1 (1) | 0 (0)
Arterial haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Chemotherapy (Cisplatin-Gemcitabine) (N=48) | Radiation: SIRT + Chemotherapy (Cisplatin-Gemcitabine) (N=41)
Anaemia (Blood and lymphatic system disorders) | 31 | 24
Leukopenia (Blood and lymphatic system disorders) | 2 | 3
Neutropenia (Blood and lymphatic system disorders) | 8 | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 7 | 8
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 3 | 0
Palpitations (Cardiac disorders) | 3 | 0
Hypoacusis (Ear and labyrinth disorders) | 6 | 4
Tinnitus (Ear and labyrinth disorders) | 5 | 5
Abdominal pain (Gastrointestinal disorders) | 10 | 11
Abdominal pain upper (Gastrointestinal disorders) | 10 | 11
Ascites (Gastrointestinal disorders) | 4 | 6
Constipation (Gastrointestinal disorders) | 24 | 18
Diarrhoea (Gastrointestinal disorders) | 15 | 10
Dry mouth (Gastrointestinal disorders) | 2 | 6
Gastric ulcer (Gastrointestinal disorders) | 0 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 3
Nausea (Gastrointestinal disorders) | 23 | 26
Stomatitis (Gastrointestinal disorders) | 8 | 9
Vomiting (Gastrointestinal disorders) | 12 | 19
Asthenia (General disorders) | 6 | 2
Fatigue (General disorders) | 34 | 32
Influenza like illness (General disorders) | 6 | 3
Oedema peripheral (General disorders) | 12 | 14
Pain (General disorders) | 6 | 4
Pyrexia (General disorders) | 6 | 10
Bronchitis (Infections and infestations) | 6 | 2
Nasopharyngitis (Infections and infestations) | 3 | 1
Alanine aminotransferase increased (Investigations) | 1 | 4
Aspartate aminotransferase increased (Investigations) | 2 | 4
Blood alkaline phosphatase increase (Investigations) | 3 | 1
Blood creatine increased (Investigations) | 4 | 3
Gamma-glutamyltransferase increased (Investigations) | 3 | 4
Neutrophil count decreased (Investigations) | 17 | 26
Platelet count decreased (Investigations) | 11 | 18
Weight decreased (Investigations) | 3 | 5
White blood cell count decreased (Investigations) | 3 | 8
Decreased appetite (Metabolism and nutrition disorders) | 16 | 24
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 3
Arthralagia (Musculoskeletal and connective tissue disorders) | 5 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 10
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 0
Dysgeusia (Nervous system disorders) | 8 | 6
Headache (Nervous system disorders) | 5 | 3
Lethargy (Nervous system disorders) | 2 | 3
Neuropathy peripheral (Nervous system disorders) | 4 | 3
Paraesthesia (Nervous system disorders) | 2 | 3
Peripheral motor neuropathy (Nervous system disorders) | 4 | 5
Peripheral sensory neuropathy (Nervous system disorders) | 14 | 9
Anxiety (Psychiatric disorders) | 3 | 2
Insomnia (Psychiatric disorders) | 4 | 5
Chronic kidney disease (Renal and urinary disorders) | 3 | 1
Renal failure (Renal and urinary disorders) | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15 | 15
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 13 | 13
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 5 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 3
Rash (Skin and subcutaneous tissue disorders) | 3 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 | 3
Embolism (Vascular disorders) | 3 | 4
Hypertension (Vascular disorders) | 7 | 7

LIMITATIONS AND CAVEATS:
SIRCCA enrollment from February 2017 (180 planned) was slow and thus enrollment terminated early in October 2019 (89 treated). Follow-up until 29 April 2021 was to ensure ≥18 months of data although the primary endpoint was underpowered. An audit to the clinical database detected issues leading to a low level of confidence in the trustworthiness of the collected data. Pharmacovigilance case reconciliation was thus also confounded. The results posted cannot be relied upon as accurate.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI must provide a proposed publication to Sponsor >=30 days prior to publication submission for review and comment on the appropriateness of the data analysis and presentation, confidential Information, and rights regarding inventions or other intellectual property. The Sponsor may extend the review period by +30 days. Publication can be delayed by Sponsor to file patent applications but such delay shall not exceed 24 months from the date of such notice to the Investigator.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-12): https://cdn.clinicaltrials.gov/large-docs/81/NCT02807181/Prot_SAP_000.pdf